CLINICAL TRIAL: NCT04975867
Title: Targeted Temperature Management Combined With Hyperbaric Oxygen Therapy in Acute Severe Carbon Monoxide Poisoning: Multicenter Randomized Controlled Clinical Trial (TTM-COHB Trial)
Brief Title: Adjunct Targeted Temperature Management in Acute Severe Carbon Monoxide Poisoning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTM-COHB trial; CR220011 (Other: Wonju Severance Christian Hospital); 2021-04-043 (Other: Inha University Hospital)
Record Dates: First submitted 2021-07-01; First posted 2021-07-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: Carbon Monoxide Poisoning; Neurologic Sequelae; Hypothermia
MeSH Terms: conditions — Carbon Monoxide Poisoning; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors of neurocognitive outcomes at 1 and 6 months after CO exposure will be blinded to the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypothermia group (Experimental): Hypothermia group is then performed at a body temperature of 33±0.5 °C during 24 h using a surface cooling device as soon as possible after the HBO and research consent. After therapeutic hypothermia ended, rewarming is done slowly between 0.2℃ - 0.5℃/h for 12 hours. After rewarming, it will be held at 36.5 ℃ for 36 hours.
  Interventions: Other: Targeted therapeutic hypothermia
- Normothermia group (Active Comparator): For normothermia group, it will be held at 36.5±0.5 ℃ for 72 hours using a surface cooling device after the HBO and research consent.
  Interventions: Other: Targeted therapeutic normothermia

INTERVENTIONS:
Other: Targeted therapeutic hypothermia — Targeted therapeutic hypothermia is then performed at a body temperature of 33±0.5 °C during 24 h using a surface cooling device as soon as possible after the HBO and research consent. After TH ended, rewarming is done slowly between 0.2℃ - 0.5℃/h for 12 hours. After rewarming, it will be held at 36.5 ℃ for 36 hours.
  Arms: Hypothermia group
Other: Targeted therapeutic normothermia — Targeted therapeutic normothermia will be held at 36.5±0.5 ℃ for 72 hours using a surface cooling device after the HBO and research consent.
  Arms: Normothermia group

SUMMARY:
This randomized trial will investigate important neurocognitive clinical outcomes of patients with acute severe carbon monoxide poisoning (ASCOP) randomized to receive either therapeutic hypothermia or normothermia combined with hyperbaric oxygen therapy (HBO).

DETAILED DESCRIPTION:
CO-poisoned patients are identified by medical history and carboxyhemoglobin (CO-Hb) value >5% (>10% in smokers). Patients presenting with acute CO poisoning will receive one HBO. ASCOP is defined as mental status showing response to painful stimulus or unresponsiveness requiring intubation for airway protection and ventilation support at the emerency department, and persistence of depressed mental status despite the HBO. After HBO treatment, eligible patients who provide consent will be randomly allocated to receive hypothermia, or normothermia treatment administered in a open label fashion except for blinding of outcome assessor.

Outcome measures will be administered at 1 month and 6 months after CO exposure. In addition, we will examine the differences in serum markers and mortality between the hypothermia and normothermia groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years.
* Patients who received HBO within 24 hours for acute CO poisoning.
* Patients who meet the definition of ASCOP (Patients incapable verbal obey after HBO).
* Signed informed consent prior to study entry.

Exclusion Criteria:

* Cardiac arrest before HBO
* Previous neurocognitive disorders
* Life-threatening underlying disease (ex: advanced cancer)
* Evidence of co-ingestion of sedative or hypnotics confirmed by intravenous flumazenil administration or history taking at the emergency department
* Absolute contraindication for TH (active severe bleeding and profound shock not controlled by vasoactive drugs)
* No admission
* The significant co-ingested drug levels, which are alter the consciousness, is confirmed from the drug analysis lab
* Pregnancy
* Burns
* More than moderate burn or Inhalation burn
* Burns complicated by other trauma
* Electrical burn
* Burns in high risk patients (Patients with chronic underlying diseases (i.e DM, ESRD, liver cirrhosis, etc) which may cause delays or aggravate the wound healing)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Main neurocognitive outcome | At 6 months after CO poisoning
  Global Deterioration Scale [range 1 - 7 (worst score)]

SECONDARY OUTCOMES:
Neurocognitive outcome | At 1 month after CO poisoning
  Global Deterioration Scale [range 1 - 7 (worst score)]
Cerebral Performance Category | At 1 month and 6 months after CO poisoning
  Cerebral Performance Category [range 1 - 5 (worst score)]
modified Rankin scale | At 1 month and 6 months after CO poisoning
  modified Rankin scale [range 0 - 6 (worst score)]
Glasgow outcome scale | At 1 month and 6 months after CO poisoning
  Glasgow outcome scale [range 1 (worst score) - 5]
mini-mental status exam | At 1 month and 6 months after CO poisoning
  mini-mental status exam
Korean version of the Modified Barthel Index | At 1 month and 6 months after CO poisoning
  Korean version of the Modified Barthel Index
Mortality in intensive care unit | Through study completion, an average of 6 months
  Number of participants with mortality in intensive care unit
Mortality in intensive care unit | Through study completion, an average of 6 months
  Rate of participants with mortality in intensive care unit
In-hospital mortality | Through study completion, an average of 6 months
  Number of participants with in-hospital mortality
In-hospital mortality | Through study completion, an average of 6 months
  Rate of participants with in-hospital mortality
Mortality | At 1, 3, and 6 months after CO poisoning
  Number of participants with all cause mortality
Mortality | At 1, 3, and 6 months after CO poisoning
  Rate of participants with all cause mortality
Length of stay in intensive care unit and hospital | Through study completion, an average of 6 months
  Length of stay in intensive care unit and hospital
Pneumonia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with the diagnosis of pneumonia. Diagnosis is established when the following two criteria are met: 1) the appearance of a new infiltrate or consolidation on chest x-ray; and 2) leukocytosis, or leukopenia, or the significant presence of meaningful bacteria in a sputum culture with the absence of other infections.
Pneumonia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with the diagnosis of pneumonia. Diagnosis is established when the following two criteria are met: 1) the appearance of a new infiltrate or consolidation on chest x-ray; and 2) leukocytosis, or leukopenia, or the significant presence of meaningful bacteria in a sputum culture with the absence of other infections.
Shock | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with shock. Diagnosis is diagnosed when a vasopressor is needed to resuscitate the patient and lactate levels exceeded 2.0 mmol/L.
Shock | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with shock. Diagnosis is diagnosed when a vasopressor is needed to resuscitate the patient and lactate levels exceeded 2.0 mmol/L.
Bradycardia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with dropped heart rate indicated drug or interventions
Bradycardia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with dropped heart rate indicated drug or interventions
Hypokalemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with serum K concentration <3.0 - 2.5 mmol/L
Hypokalemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with serum K concentration <3.0 - 2.5 mmol/L
Hyperkalemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with serum K concentration >6.0 - 7.0 mmol/L
Hyperkalemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with serum K concentration >6.0 - 7.0 mmol/L
Hyperglycemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with change (Insulin therapy initiated) in daily management from baseline for serum glucose
Hyperglycemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with change (Insulin therapy initiated) in daily management from baseline for serum glucose
Hypophosphatemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with a disorder characterized by laboratory test results that indicate a low concentration of phosphates in the blood and indicated replacement therapy
Hypophosphatemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with a disorder characterized by laboratory test results that indicate a low concentration of phosphates in the blood and indicated replacement therapy
Hypomagnesemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with serum magnesium <0.9 - 0.7 mg/dL
Hypomagnesemia | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with serum magnesium <0.9 - 0.7 mg/dL
Prolonged prothrombin Time International Normalized Ratio | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with >2.5 x upper limit of the normal range and bleeding
Prolonged prothrombin Time International Normalized Ratio | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with >2.5 x upper limit of the normal range and bleeding
Prolonged activated partial thromboplastin time | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Number of participants with >2.5 x upper limit of the normal range and bleeding
Prolonged activated partial thromboplastin time | During the intervention (therapeutic hypothermia or normothermia) period (72 hours)
  Rate of participants with >2.5 x upper limit of the normal range and bleeding
S100ß (serum) | Within 14 days after CO exposure
  Concentration of S100ß (serum)
Neuronal specific enolase (serum) | Within 14 days after CO exposure
  Concentration of neuronal specific enolase (serum)
Brain magnetic resonance image (MRI) | Within 14 days after CO exposure
  Number of participants with brain injury in brain MRI
Brain magnetic resonance image (MRI) | Within 14 days after CO exposure
  Rate of participants with brain injury in brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sung Cha, MD, Principal Investigator — Wonju Severance Christian Hospital
Locations (2):
- South Korea (2):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inha University Hospital, Incheon, Incheon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SJ, Thom SR, Kim H, Hwang SO, Lee Y, Park EJ, Lee SJ, Cha YS. Effects of Adjunctive Therapeutic Hypothermia Combined With Hyperbaric Oxygen Therapy in Acute Severe Carbon Monoxide Poisoning. Crit Care Med. 2020 Aug;48(8):e706-e714. doi: 10.1097/CCM.0000000000004419. PMID 32697512